CLINICAL TRIAL: NCT03671200
Title: Correlation Between Caries Experience in Primary Molars and First Permanent Molars Among a Group of Egyptian Children: A Cross Sectional Study
Brief Title: Correlation Between Caries Experience in Primary Molars and First Permanent Molars
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, dema abdulhameed theyab, Principal investigator, Cairo University
Other Study IDs: CEBD-CU-2018-08-10
Record Dates: First submitted 2018-09-08; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Caries,Dental
Keywords: Primary teeth; Permanent first molar; Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross- sectional observational study which will investigate whether data of past caries experience of the primary molars of 6-9 years old children can serve as an indicator for caries development in first permanent molars.as the first permanent molars is selected to represent the future caries status of the permanent dentition.

DETAILED DESCRIPTION:
Study Design:

A cross sectional study to investigate if there is any correlation between caries experience in primary molars and first permanent molars among a group of Egyptian children. All the procedures will be explained to the parents or guardians prior to the investigation.An informed consent will be signed by the parents Study design: cross sectional study design. Data for this particular study will be collected from the clinic of Pediatric Dentistry and dental public health Department, Faculty of Dentistry, Cairo University.

Methods Clinical examination will be carried out while the child is sitting on dental unit, using sterile diagnostic set (mirror and explorer) in daylight. No diagnostic radiographs will be taken.

A custom-made examination chart will be filled for each child including date, name, age, address, gender, medical history and previous dental treatment. Parents data includes: level of education and oral hygiene level.

Prior to performing dental examination, the child will be asked to rinse his mouth with tap water and the teeth will be cleaned with sterile cotton.

The examiner will carefully inspect all surfaces of the teeth, for proper diagnosis, the teeth were dried thoroughly with an air syringe. It will be important to see clearly and to use the air syringe to distinguish readily cervical or interproximal caries.

All the primary teeth will be evaluated using deft index and permanent teeth will be evaluated using DMF index, both according to WHO criteria.

(WHO, 2003) criteria: Clinical caries lesion shows the following criteria

Lesion in pit or fissure, or on a smooth tooth surface with cavitated undermined enamel, or a detectably softened floor or wall.

Teeth with recurrent dental caries. In cases where the crown has been destroyed by caries and only the root is left, the caries is judged to be crown caries.

Lesions not considered as clinical dental caries White or chalky spots (early carious lesion). Stained enamel pits or fissures without visible cavitation or soft floor or walls during examination by sharp explorer.

Dark, shiny, hard, pitted areas of enamel in a tooth showing signs of moderate to severe enamel fluorosis.

Each child and parents will be given two printed sheet translated into Arabic, after the end of the diagnosis, which will include his/her caries status, the right oral hygiene method to be followed in order to maintain a good oral health status and any caries lesions that need treatment by restorative material or preventive measures

ELIGIBILITY:
Inclusion Criteria:

1. Children ages from six to nine years
2. Both sexes.
3. Parent and children cooperation.
4. Healthy children.
5. Children with sound and carious primary molars and erupted all of the first permanent molars.

Exclusion Criteria:

1. Children age under 6 or more than 9 years.
2. Children had a complex metabolic or medical disorder.
3. Parents that will not sign the consent.
4. Children with missing or unerupted first permanent molars.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A convenient of Egyptian children aged 6-9 years attending the clinic of Pediatric Dentistry and dental public health Department, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
decay extracted filled primary teeth index (deft index) | Data collection will be performed within one year from the starting date of the study.
  caries experience in primary molars. Clinical examination will be performed at once for each patient, the examination will be done in the clinic using an explorer and mirror after drying the teeth to detect the presence of caries in the upper and lower primary molars.
decayed missing filled permanent teeth (DMFT index) | Data collection will be performed within one year from the starting date of the study.
  Caries experience in first permanent molars.Clinical examination will be performed at once for each patient, the examination will be done in the clinic using an explorer and mirror after drying the teeth to detect the presence of caries in the upper and lower permanent first molars.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03671200/Prot_000.pdf